CLINICAL TRIAL: NCT02798640
Title: A Single Center Prospective Comparative Study to Evaluate the Performance of a Upper Torso Garment Containing 100% Celliant Fibers That Emits Far Infrared (FIR) From Ceramic Particles Contained Within the Fibers in Healthy Subjects
Brief Title: Comparative Study Evaluating Performance of Celliant Fibers on Tissue Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristopher Washington (Industry)
Responsible Party: Sponsor-Investigator, Kristopher Washington, Study Coordinator, Hologenix, LLC
Organization: Hologenix, LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HC1-2
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Transcutaneous Oxygen Tension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Subject wearing Celliant garment
  Interventions: Device: Celliant
- Control (Placebo Comparator): Subject wearing non-celliant control garment
  Interventions: Device: Control

INTERVENTIONS:
Device: Celliant — 100% Celliant garment
  Arms: Active
Device: Control — Control Garment
  Arms: Control

SUMMARY:
The study will evaluate changes in transcutaneous oxygen tension (tcPO2,), and the inferred change in local cutaneous blood flow, in healthy subjects wearing a control and a 100% Celliant® fiber upper torso garment.

DETAILED DESCRIPTION:
Adequate blood supply is necessary for many physiologic processes. However, there are few valid, reproducible, non-invasive methods with which to assess it. One such measure is transcutaneous partial pressure of oxygen (tcPO2). This measurement is a non-invasive method of measuring oxygen tension at the skin surface; represents the amount of oxygen diffusing outward across the skin; and can be used as a surrogate for arterial perfusion. This method is reproducible with clinically acceptable intrasubject variability; is used for a variety of conditions, including peripheral vascular disease evaluation, predicting the outcome of patients requiring amputation and survival of skin grafts; and correlates well to angiography and increases in blood flow rates. However, tcPO2 is affected by many variables, including oxygen concentration in inspired air, lung function and hemoglobin saturation, as well as local factors, such as skin thickness, sympathetic tone, the presence of inflammation, capillary formation and skin oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than or equal to18 years of age
* Men and women between the ages of 18 and 60 years
* Able to understand and consent to the study
* Able to follow directions of the Study Coordinators and/or the Principal Investigator
* Able to complete the study
* Male or female subjects of any ethnic origin such that the balance across ages and among population groups is reflective of the site population

Exclusion Criteria:

* Active smokers
* No history of cardiovascular disease
* No history of peripheral vascular disease
* Engaged in recreational drug use for the six months prior to the start of the study
* Eaten within two (2) hours of the study
* Consumed caffeine within four (4) hours prior to the study
* Consumed alcohol with forty-eight (48) hours prior to the study
* Subjects with any unstable medical or psychiatric problem
* Subjects who are pregnant or nursing mothers
* Subjects who are currently taking part in another clinical study or have taken part in a drug or device study, in the past month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in transcutaneous oxygen tension (tcPO2) | 0,30,60,90 minutes
  comparison of individual measurements taken at these time points

SECONDARY OUTCOMES:
Changes in local skin temperature by infrared imaging | 0,30,60,90 minutes
  comparison of individual measurements taken at these time points

CONTACTS AND LOCATIONS:
Overall Officials: Ian L Gordon, M.D., Principal Investigator — University of California Medical Center Wound Clinic; Kristopher Washington, B.S., Study Director — Hologenix, LLC
Locations (1):
- Hologenix, LLC, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Informed Consent Form — https://mega.nz/#!C5U1HZwI!7XB2jar-JDElrnYOZTbwg0RD5T1WPQEv3HkzT0XPXz8
- Available data/document: Clinical Investigation plan — https://mega.nz/#!3gEnFCDK!DK911mpjGBw_bAKdfsR4F2RgzCQG7mYR3oBqrVkRtpA
- Available data/document: Clinical Study Report — https://mega.nz/#!S1tThKrL!gaWPII28P3I0BLBrLD9iZJYRqb2R1x-uZT5djgV4ML8